CLINICAL TRIAL: NCT03129997
Title: Effect of Gluten-free Diets on Anthropometric and Dietary Data of Healthy Eutrophic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Jacqueline Isaura Alvarez Leite, MD,Ph.D, Federal University of Minas Gerais
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 49480215000005149H
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: crossover double masked model
Who Masked: Participant, Investigator
Masking Description: volunteers received placebo or gluten corn muffins that are similar in taste and appearance. Investigator does not know who is receiving placebo or gluten muffins. During analyses, each sample is coded to avoid volunteer or phase identification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluten test food (Active Comparator): volunteers will receive 2 corn based muffins containing 7,5g of gluten/muffin to be consumed daily for 3 weeks
  Interventions: Dietary Supplement: Gluten test food
- Placebo test food (Placebo Comparator): volunteers will receive 2 corn based muffins to be consumed daily in any meal for 3 weeks
  Interventions: Dietary Supplement: Gluten test food

INTERVENTIONS:
Dietary Supplement: Gluten test food — Dietary supplement: corn muffins with 7.5g of gluten/muffin Two muffin were blindly administered for 21 days

SUMMARY:
The objective is to evaluate, in healthy, eutrophic women, if gluten intake influences on body weight, basal metabolic rate and macronutrient intake. In a crossover double masked model, 30 volunteers will be randomized into two groups, half of them will initiate the experiment by taking 2 "placebo" muffins daily for 3 weeks (Placebo phase) and the remnant volunteers will take 2 "gluten" muffins for 3 weeks (Gluten phase). After one day of wash out, the volunteers will be transferred for the other phase to complete 3 more experimental weeks.

DETAILED DESCRIPTION:
The objective is to evaluate in eutrophic women the impact of intake of moderate amounts of wheat gluten on body weight basal metabolic rate and possible relation to macronutrient intake. For this, 30 volunteers will kept on a restricted diet in gluten-free foods of 6 weeks. At the first moment, a structured Food Frequency Questionnaire will be applied, as well as a 24-hour food register, to evaluate the average food and gluten daily intake. The volunteers will be randomized into two groups, half of them will initiate the experiment by taking 2 placebo muffins daily for 3 weeks (Placebo phase) and the remnant volunteers will take 2 gluten muffins for 3 weeks (Gluten phase). After one day of wash out, the volunteers will be transferred for the other phase to complete 3 more experimental weeks. During these 6 experimental weeks, all volunteers will be instructed to exclude any food containing gluten from their diet. The test food (gluten and placebo muffins) will be produced in the Laboratory of Dietetic Technique of the School of Nursing of the Federal University of Minas Gerais and delivered weekly to each volunteer. Placebo test foods is a corn-based muffin of about 45g. In the Gluten muffins, 10g of corn is replaced by 10g of gluten (corresponding to 7.5g of gluten protein). Each volunteer will be instructed to take 2 (placebo or gluten) muffin/day. To evaluate diet adherence and signs and symptoms of intolerances, volunteers will fill a questionnaire weekly, informing about the consumption of the test food, eventual intake of food containing gluten, and the presence of gastrointestinal signs and symptoms such as constipation, diarrhea, nausea or vomiting etc.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 40
* Body Mass Index (BMI) between 18.5 and 24.9 kg / m²
* Sign of informed consent
* Absence of associated chronic diseases

Exclusion Criteria:

* Postmenopausal patients
* Onset of chronic medication
* discontinuance of test food intake for 2or more days
* Do not attend 2 of the 3 meetings.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Changes in body Weight | 1st, 3rd and 6th weeks
  measured in scale presented in kg

SECONDARY OUTCOMES:
Changes in resting metabolic rate | 1st, 3rd and 6th weeks
  measured by indirect calorimetry in kcal/kg or kcal/day
Changes in macronutrient intake | 1st, 3rd and 6th weeks
  calculation of food intake based on 24h diary - result in % kcal
waist circumference | 1st, 3rd and 6th weeks
  measured in cm
Height | 1st week
  measured in meters
BMI | 1st, 3rd and 6th weeks
  calculated by body weigh / square of height

CONTACTS AND LOCATIONS:
Overall Officials: JAQUELINE I ALVAREZ-LEITE, Principal Investigator — Federal University of Minas Gerais

IPD SHARING:
Plan to Share IPD: No